CLINICAL TRIAL: NCT02389647
Title: Identification of Novel Molecular Markers for Cerebral Ischemia From Patients With Minor and Devastating Ischemic Injury
Status: Completed | Type: Observational
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: Translational Genomics Research Institute (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Norissa Honea, Research clinician, St. Joseph's Hospital and Medical Center, Phoenix
Other Study IDs: 13BN094; 5UH2TR000891 (NIH)
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Cerebral Ischemia
MeSH Terms: conditions — Brain Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Endovascular group: Subjects undergoing elective endovascular catheterization for coiling of unruptured cerebral aneurysms. Four blood draws of 5mL each: (1) prior to initiation of procedure; (2) at the time of catheterization of major cerebral vessels, (3) immediately after the procedure, and (4) 24-hours after the procedure.
- Ischemic stroke group: Subjects who present to the emergency department with ischemic infarcts of <6 hours. Four blood draws of 5mL each: (1) at time of enrollment but prior to tPA, (2) 6 hours post-tPA, (3) 12 hours post-tPA, and (4) 24 hours post-tPA.
- Intracranial hemorrhage: Subjects who present to the emergency department with intracranial hemorrhage. One 5mL blood draw within 24 hours of onset.

SUMMARY:
The purpose of this study is to use an iatrogenic model of stroke, meaning those strokes inadvertently caused by endovascular coiling of elective aneurysms, to study the biology of stroke in humans.

DETAILED DESCRIPTION:
Ischemic stroke is one of the top causes of morbidity and mortality in the United States. Despite a great deal of effort to improve outcomes of patients with ischemic cerebral strokes, the lack of a bona fide animal model representative of cerebral ischemia in man makes the study of the pathological processes involved difficult. Additionally, the subtle but significant differences between biology of animal models and the biology of humans make translatability of animal results to humans difficult.

The purpose of this study is to use an iatrogenic model of stroke, meaning those strokes inadvertently caused by endovascular coiling of elective aneurysms, to study the biology of stroke in humans. Clinical evidence suggests that simple catheterization of cerebral vasculature causes small, usually clinically silent, embolic strokes. These strokes are evident on MRI scans. Additionally, since the practitioner knows the onset of an interventional procedure, he by default knows the timing of injury. This simple model allows one to study stroke in real-time with knowledge of the time of onset. Magnetic resonance imaging (MRI) evaluation allows the practitioner to identify the volume of stroke caused by the intervention. Alternatively, patients who present to the emergency room with large ischemic infarcts provide a natural control population for this study. These patients present with large, usually devastating strokes. In most cases the timing of the onset of deficit is known. The investigators propose to use the simple model of ischemia from endovascular interventions with the more obvious devastating cases of ischemic stroke who present to the emergency room to better understand the molecular pathways involved in stroke.

Rationale: Global analysis of biological markers is an established mechanism to study complex disease processes. The introduction of microarray technology and systems wide analysis has improved the understanding of various biological and disease processes. This revolution has been ongoing since the early 1990's. The rationale for performing these studies is to augment the understanding of the basic mechanisms of stroke in humans. As previously mentioned, there is no bona fide model of stroke and the researchers' experimental design provides a rather simple in human model for cerebral ischemia.

The study requires four blood draws, each 5 mL in volume; blood draws are timed with normal times of blood draw these patients would be experiencing and do not place the patient at any additional risk.

The blood samples will be analyzed as follows: total ribonucleic acid (RNA), including the microRNA fraction, and protein will be isolated and quantified from the blood samples. The researchers will load the RNA samples onto Febit microRNA arrays. The Febit miRNA chip has all of the known human miRNAs and miRNA star sequences from Sanger's miRBase 14. With this platform total RNA is loaded directly onto the array. There are no RNA labeling or amplification steps. miRNA hybridization on the chip is followed by a microfluidic primer extension assay. In this case, only hybridization of the correct miRNA to the probe allows the primer extension step to proceed efficiently, giving the array high sensitivity and specificity. In addition, the researchers have created custom microarrays, adding several spike-in controls. Our spike-ins provide feedback on the variability in RNA isolation and are an additional signal for array normalization. The protein fraction will be analyzed using Ray Biotech's Quantibody Arrays. These are arrays of antibodies that are designed to capture specific protein species (the researchers will target approximately 120 unique proteins) in a fully quantitative fashion. These arrays essentially function as the traditional enzyme-linked immunosorbent assay (ELISA) but on a glass slide substrate. The assays offer several advantages over ELISA's, including the requirement for very low amounts of sample input but, perhaps more importantly, they facilitate the quantitative investigation of hundreds of proteins at once and therefore greatly accelerate the ability to search for and identify protein-based signatures and/or biomarkers. The data will be statistically analyzed using statistical tools that are deemed appropriate at the time of data analysis by investigators from TGen and Dr. Kalani. Drs. Kalani and Nakaji will then correlate the identity and quantity of identified molecular markers, their temporal appearance, concentration, and disappearance to the collected clinical data.

A neuroradiologist will perform evaluation and interpretation of the computerized axial tomography (CT)/MRI scans collected during the subject's inpatient stay and outpatient visits. The neuroradiologist will be recording size and caliber of the blood vessels, looking for malformations, dissections, aneurysms, or other abnormalities.

The researchers will also correlate the level of identified markers to how well the patient performs upon discharge from the hospital and at followup for up to two years from discharge, using Modified Rankin Scale scores and Glasgow Outcome Scale (GOS). As a part of followup, researcher will assess time to return to work (if applicable), complaints, results of followup laboratory (complete blood counts, coagulation studies, response to anti-platelet medications including aspirin resistance assay and the p2yp12 assays, and basic metabolic panels) and imaging, and an updated complete history and physical to identify new conditions that may have resulted post-ischemia. This information will be collected at the time of followup with the neurosurgeons. Once this is done, if a candidate microRNA or protein is identified, the researchers will share the results (again in a manner that excludes any patient specific information) with our collaborators (Department of Health and Human Services associated organizations such as the NIH).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who present with ischemic infarcts to the emergency department with a known time of infarct.
* Time of infarct <6 hours.
* Adult patients with unruptured aneurysms who present for elective endovascular coiling of the aneurysm(s).

Exclusion Criteria:

* Under 18 years of age.
* Patients arriving to the emergency department >6 hours after infarct.
* Patients considered as not candidates for further care.
* Patients with ruptured cerebral aneurysm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects presenting to facility and diagnosed with ischemic stroke, intracranial hemorrhage, or elective endovascular coiling of unruptured aneurysm.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-03; Primary Completion 2019-10-24 (Actual); Study Completion 2019-10-24 (Actual)

PRIMARY OUTCOMES:
Identification of biomarkers selective for ischemia of the central nervous system | After each blood draw

CONTACTS AND LOCATIONS:
Overall Officials: Peter Nakaji, MD, Principal Investigator — Saint Joseph's Hospital and Medical Center/Barrow Neurological Institute
Locations (1):
- St. Joseph's Hospital and Medical Center/Barrow Neurological Institute, Phoenix, Arizona, United States